CLINICAL TRIAL: NCT00264810
Title: RNS® System Pivotal-A Clinical Investigation
Brief Title: RNS® System Pivotal Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NeuroPace (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP10004
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Epilepsy
Keywords: Responsive Stimulation; Brain Stimulator; Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (stimulation ON) (Active Comparator): Group of subjects that have undergone RNS® System implantation that are randomized to receive RNS® System responsive stimulation (i.e. responsive stimulation enabled or turned ON) during the Blinded Evaluation Period. Stimulation is enabled during the Stimulation Optimization Period (second month post-implant) and may continue throughout the subject's participation in the study.
  Interventions: Procedure: RNS® System implantation; Device: RNS® System responsive stimulation
- Sham Group (stimulation OFF) (Sham Comparator): Group of subjects that have undergone RNS® System implantation that are randomized to receive sham-stimulation (i.e. responsive stimulation disabled or turned OFF) during the Blinded Evaluation Period. Stimulation is enabled after transition into the Open Label Period (sixth month post-implant) and may continue for the remainder of the subject's participation in the study.
  Interventions: Procedure: RNS® System implantation

INTERVENTIONS:
Procedure: RNS® System implantation — Using standard neurosurgical techniques the surgical team implants the RNS® System, which includes the RNS® Neurostimulator and intracranial NeuroPace® Leads. Up to 4 Leads (Cortical Strips and/or Depth Leads) are placed in or near the epileptogenic focus/foci. The Neurostimulator is placed in the skull and connected to up to 2 Leads. At first the Neurostimulator is programmed to record brain activity (electrographic patterns). The neurologist or neurosurgeon reviews the recorded electrographic patterns and identifies abnormal (epileptiform, or seizure-like) activity. The Neurostimulator is then programmed to detect the abnormal activity.
Device: RNS® System responsive stimulation — The RNS® System is programmed to provide responsive stimulation (stimulation is ON or enabled). Upon detecting electrographic patterns, previously identified by the neurologist or neurosurgeon as abnormal (epileptiform, or seizure-like) activity, the Neurostimulator provides brief pulses of electrical stimulation through the Leads to interrupt those patterns. The typical patient is treated with a cumulative total of 5 minutes of stimulation a day.
  Arms: Treatment Group (stimulation ON)

SUMMARY:
The RNS® System Pivotal study is designed to assess safety and demonstrate that the RNS® System is effective as an adjunctive (add-on) therapy in reducing the frequency of seizures in individuals 18 years of age or older with partial onset seizures from no more than two foci (two areas of the brain) that are refractory (drug-resistant or hard-to-treat) to two or more antiepileptic medications. Patients continue to receive their epilepsy medications while participating in the study.

DETAILED DESCRIPTION:
NeuroPace, Inc. is sponsoring an investigational device study of the RNS® System, the first closed loop responsive brain stimulator designed to treat refractory epilepsy. The RNS® System Pivotal study is a multi-center, randomized, double-blinded, sham-stimulation controlled investigation being conducted at 32 epilepsy centers throughout the United States. The study is designed to assess safety and demonstrate that the RNS® System is effective in reducing the frequency of medically uncontrolled and disabling partial onset seizures that start from one or two areas of the brain.

The RNS® Neurostimulator (a pacemaker-like device) and NeuroPace® Leads (tiny wires with electrodes) are implanted in the head. The Neurostimulator is a battery powered, microprocessor controlled device that detects and stores records of electrographic patterns (such as epileptiform, or seizure-like, activity) from the Leads within the brain. When the device detects an electrographic pattern, it responds by sending electrical stimulation through the Leads to a small part of the patient's brain to interrupt the electrographic pattern. This type of treatment is called responsive stimulation, but it is not yet known if it will work for the treatment of epilepsy. Direct brain stimulation therapy has already received approval in the United States, Europe, Canada, and Australia for the treatment of Essential Tremor and Parkinson's disease. Direct brain stimulation is not approved for the treatment of epilepsy.

Subjects participating in the RNS® System Pivotal study must met inclusion criteria, including localization of epileptogenic region(s), prior to enrolling in the study. Throughout the entire study, subjects or their caregivers must keep a seizure diary. Seizure frequency, seizure severity, and antiepileptic medications, as well as physical and emotional health will be monitored and recorded throughout the study.

Upon demonstrating the required seizure frequency and stable antiepileptic medications over 3 consecutive months of the Baseline (pre-implant) Period, subjects will qualify for RNS® System implantation. Antiepileptic medications should continue to remain stable until 6 months post-implant. The surgical procedure will be performed within one month of qualification.

The RNS® Neurostimulator is cranially implanted and connected to one or two NeuroPace® Leads implanted in the brain. The investigational team will determine the placement of the Leads based on prior localization of the epileptogenic region, according to standard localization procedures. Detection of epileptiform activity will be enabled for all subjects during the 1 month Post-Operative Stabilization Period. Subjects will be randomized 1:1 to either the Treatment or Sham group prior to starting the 1 month Stimulation Optimization Period. During this period subjects are seen on a weekly basis by the Treatment Protocol investigator. Responsive stimulation will be enabled and optimized for subjects randomized to the Treatment group. Subjects randomized to the Sham group will be seen for simulated stimulation programming in order to maintain the treatment blind.

The Blinded Evaluation Period is comprised of months 3, 4, and 5 post-implant. Subjects in the Treatment group will receive responsive stimulation and subjects in the Sham group will not. Subjects will not know whether responsive stimulation is being delivered or not. At the end of the 5th month, all subjects' transition into the Open Label Evaluation Period during which all subjects may receive responsive stimulation and antiepileptic medications may be adjusted as medically required.

Subjects will be followed for 2 years post-implant. Throughout study participation, both effectiveness and safety data will be monitored continuously, and reviewed and documented by the study investigator at study appointments scheduled every month for the first year post-implant, then every 3 months.

ELIGIBILITY:
Inclusion Criteria for enrollment:

1. Subject has disabling motor simple partial seizures, complex partial seizures, and/or secondarily generalized seizures. Disabling refers to seizures that are severe enough to cause injuries or significantly impair functional ability.
2. Subject's seizures are distinct, stereotypical events that can be reliably counted.
3. Subject failed treatment with a minimum of 2 anti-seizure medications.
4. Subject has remained on the same antiepileptic medication(s) over the 3 most recent consecutive months (other than acute, intermittent use of benzodiazepines). Subjects on the ketogenic diet are permitted if the diet has been stable for the preceding 3 months.
5. Subject reports having an average of 3 or more disabling motor simple partial seizures, complex partial seizures and/or secondarily generalized seizures per month over the 3 most recent consecutive months, with no month with less than 2 seizures.
6. Subject is between the ages of 18 and 70 years.
7. Subject has undergone diagnostic testing that has identified no more than 2 epileptogenic regions.
8. Subject is male or a female of childbearing potential using a reliable method of contraception or is at least two years post-menopause.
9. Subject or legal guardian is able to provide appropriate consent to participate.
10. Subject can be reasonably expected to maintain a seizure diary alone or with the assistance of a competent individual.
11. Subject is able to complete regular office and telephone appointments per the protocol requirements.
12. Subject is willing to be implanted with the RNS® System as a treatment for his/her seizures.
13. Subject is able to tolerate a neurosurgical procedure.
14. Subject is considered a good candidate to be implanted with the RNS® System.

Note: A subject is still eligible to participate if antiepileptic medication(s) were temporarily discontinued for the purposes of diagnostic or medical procedures during the preceding 3 months.

Exclusion Criteria for enrollment:

1. Subject has been diagnosed with psychogenic or non-epileptic seizures in the preceding year
2. Subject has been diagnosed with primarily generalized seizures.
3. Subject has experienced unprovoked status epilepticus in the preceding year.
4. Subject has a clinically significant or unstable medical condition (including alcohol and/or drug abuse) or a progressive central nervous system disease.
5. Subject is taking chronic anticoagulants.
6. Subject has been diagnosed with active psychosis, major depression or suicidal ideation in the preceding year. Subjects with post-ictal psychiatric symptoms need not be excluded.
7. Subject is pregnant or planning on becoming pregnant in the next 2 years.
8. Subject is enrolled in a therapeutic investigational drug or device trial.
9. Subject has an implanted Vagus Nerve Stimulator (VNS) or is unwilling to have the VNS explanted. (VNS therapy must have been discontinued for at least 3 months prior to enrollment.)
10. Subject has had therapeutic surgery to treat epilepsy in the preceding 6 months.
11. Subject has had a cranial neurosurgical procedure (including endovascular procedures) other than an epilepsy surgery involving the skull or brain in the previous month.
12. Subject is implanted with an electronic medical device that delivers electrical energy to the head.
13. Subject is an unsuitable candidate for neurosurgery.
14. Subject requires repeat MRIs in which the head is exposed to the radio frequency field.
15. Subject's epileptogenic region(s) is/are located caudal to the level of the thalamus.
16. Implantation of the RNS® Neurostimulator and Lead(s) would present unacceptable risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Barkley, MD, Principal Investigator — Johns Hopkins University; Michel Berg, MD, Principal Investigator — University of Rochester; Gregory Bergey, MD, Principal Investigator — Henry Ford Hospital; Carl Bazil, MD, Principal Investigator — Columbia University / Columbia Presbyterian Medical Center; Andrew Cole, MD, Principal Investigator — Massachusetts General Hospital; Michael Duchowny, MD, Principal Investigator — Nicklaus Children's Hospital f/k/a Miami Children's Hospital; Robert Duckrow, MD, Principal Investigator — Yale University; Jonathan Edwards, MD, Principal Investigator — Medical University of South Carolina; Stephan Eisenschenk, MD, Principal Investigator — University of Florida at Gainesville; A. James Fessler, MD, Principal Investigator — University of Rochester; Nathan Fountain, MD, Principal Investigator — University of Virginia; Eric Geller, MD, Principal Investigator — St. Barnabas Medical Center; Robert Gross, MD, Principal Investigator — Emory University; Ryder Gwinn, MD, Principal Investigator — Swedish Medical Center; Christianne Heck, MD, Principal Investigator — University of Southern California; Barbara Jobst, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; David King-Stephens, MD, Principal Investigator — California Pacific Medical Center; James Leiphart, MD, Principal Investigator — George Washington University; W. Richard Marsh, MD, Principal Investigator — Mayo Clinic; Andrew Massey, MD, Principal Investigator — Via Christi Comprehensive Epilepsy Center; Eli Mizrahi, MD, Principal Investigator — Baylor College of Medicine; Dileep Nair, MD, Principal Investigator — The Cleveland Clinic; Cormac O'Donovan, MD, Principal Investigator — Wake Forest University Health Sciences; A. LeBron Paige, MD, Principal Investigator — University of Alabama at Birmingham; Yong Park, MD, Principal Investigator — Medical College of Georgia / Georgia Health Sciences University; Paul Rutecki, MD, Principal Investigator — University of Wisconsin, Madison; Vicenta Salanova, MD, Principal Investigator — Indiana University; Christopher Skidmore, MD, Principal Investigator — Thomas Jefferson University; Michael Smith, MD, Principal Investigator — Rush University Medical Center / Epilepsy Center; David Spencer, MD, Principal Investigator — Oregon Health and Science University; Paul Van Ness, MD, Principal Investigator — University of Texas Southwestern Medical Center; Robert Wharen, MD, Principal Investigator — Mayo Clinic; Richard Zimmerman, MD, Principal Investigator — Mayo Clinic
Locations (32):
- United States (32):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida at Gainesville, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia / Georgia Health Sciences University, Augusta, Georgia
  - Rush University Medical Center/ Epilepsy Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Via Christi Comprehensive Epilepsy Center, Wichita, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Columbia University / Columbia Presbyterian Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Background] Behrens E, Schramm J, Zentner J, Konig R. Surgical and neurological complications in a series of 708 epilepsy surgery procedures. Neurosurgery. 1997 Jul;41(1):1-9; discussion 9-10. doi: 10.1097/00006123-199707000-00004. PMID 9218289
- [Background] Beric A, Kelly PJ, Rezai A, Sterio D, Mogilner A, Zonenshayn M, Kopell B. Complications of deep brain stimulation surgery. Stereotact Funct Neurosurg. 2001;77(1-4):73-8. doi: 10.1159/000064600. PMID 12378060
- [Background] Fountas KN, Smith JR. A novel closed-loop stimulation system in the control of focal, medically refractory epilepsy. Acta Neurochir Suppl. 2007;97(Pt 2):357-62. doi: 10.1007/978-3-211-33081-4_41. PMID 17691324
- [Background] Fountas KN, Smith JR. Subdural electrode-associated complications: a 20-year experience. Stereotact Funct Neurosurg. 2007;85(6):264-72. doi: 10.1159/000107358. Epub 2007 Aug 17. PMID 17709978
- [Background] Hamer HM, Morris HH, Mascha EJ, Karafa MT, Bingaman WE, Bej MD, Burgess RC, Dinner DS, Foldvary NR, Hahn JF, Kotagal P, Najm I, Wyllie E, Luders HO. Complications of invasive video-EEG monitoring with subdural grid electrodes. Neurology. 2002 Jan 8;58(1):97-103. doi: 10.1212/wnl.58.1.97. PMID 11781412
- [Background] Hariz MI. Complications of deep brain stimulation surgery. Mov Disord. 2002;17 Suppl 3:S162-6. doi: 10.1002/mds.10159. PMID 11948772
- [Background] Joint C, Nandi D, Parkin S, Gregory R, Aziz T. Hardware-related problems of deep brain stimulation. Mov Disord. 2002;17 Suppl 3:S175-80. doi: 10.1002/mds.10161. PMID 11948774
- [Background] Koller WC, Lyons KE, Wilkinson SB, Troster AI, Pahwa R. Long-term safety and efficacy of unilateral deep brain stimulation of the thalamus in essential tremor. Mov Disord. 2001 May;16(3):464-8. doi: 10.1002/mds.1089. PMID 11391740
- [Background] Oh MY, Abosch A, Kim SH, Lang AE, Lozano AM. Long-term hardware-related complications of deep brain stimulation. Neurosurgery. 2002 Jun;50(6):1268-74; discussion 1274-6. doi: 10.1097/00006123-200206000-00017. PMID 12015845
- [Background] Tanriverdi T, Ajlan A, Poulin N, Olivier A. Morbidity in epilepsy surgery: an experience based on 2449 epilepsy surgery procedures from a single institution. J Neurosurg. 2009 Jun;110(6):1111-23. doi: 10.3171/2009.8.JNS08338. PMID 19199440
- [Background] Wong CH, Birkett J, Byth K, Dexter M, Somerville E, Gill D, Chaseling R, Fearnside M, Bleasel A. Risk factors for complications during intracranial electrode recording in presurgical evaluation of drug resistant partial epilepsy. Acta Neurochir (Wien). 2009 Jan;151(1):37-50. doi: 10.1007/s00701-008-0171-7. Epub 2009 Jan 8. PMID 19129963
- [Result] Morrell MJ; RNS System in Epilepsy Study Group. Responsive cortical stimulation for the treatment of medically intractable partial epilepsy. Neurology. 2011 Sep 27;77(13):1295-304. doi: 10.1212/WNL.0b013e3182302056. Epub 2011 Sep 14. PMID 21917777
- [Derived] Meador KJ, Kapur R, Loring DW, Kanner AM, Morrell MJ; RNS(R) System Pivotal Trial Investigators. Quality of life and mood in patients with medically intractable epilepsy treated with targeted responsive neurostimulation. Epilepsy Behav. 2015 Apr;45:242-7. doi: 10.1016/j.yebeh.2015.01.012. Epub 2015 Mar 26. PMID 25819949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Level 4 epilepsy centers, as categorized by the National Association of Epilepsy Centers (NAEC), through the United States.
Pre-assignment Details: Besides continuing to meet all I/E criteria, in order to undergo initial implant and be assigned to a group (randomized), subjects were required to maintain an average of 3 or more disabling partial seizures per month and remain on the same AED regimen (except for acute, intermittent use of benzodiazepines), for 3 consecutive months (12 weeks).
Period: Baseline
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF)
Started | 120 (Subjects were not assigned to a group until the end of the Post-Operative Stabilization Period.) | 120 (Subjects were not assigned to a group until the end of the Post-Operative Stabilization Period.)
Completed | 97 (Subjects were not assigned to a group until the end of the Post-Operative Stabilization Period.) | 94 (Subjects were not assigned to a group until the end of the Post-Operative Stabilization Period.)
Not Completed | 23 | 26
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Physician Decision | 7 | 8
Not completed — Subject Compliance Failure | 3 | 3
Not completed — Insufficient Seizure Frequency | 2 | 2
Not completed — Did not Meet/Maintain Study I/E Criteria | 1 | 2
Not completed — Other | 0 | 1
Period: Post-Operative Stabilization Period
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF)
Started | 97 (Subjects were not assigned to a group until the end of the Post-Operative Stabilization Period.) | 94 (Subjects were not assigned to a group until the end of the Post-Operative Stabilization Period.)
Completed | 97 | 94
Not Completed | 0 | 0
Period: Stimulation Optimization Period
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF)
Started | 97 | 94
Completed | 96 | 93
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1
Period: Blinded Evaluation Period
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF)
Started | 96 | 93
Completed | 95 | 92
Not Completed | 1 | 1
Not completed — Explant due to infection | 1 | 1
Period: Open Label Evaluation Period
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF)
Started | 95 | 92
1-year Post-implant | 92 | 90
Completed | 89 | 86
Not Completed | 6 | 6
Not completed — Explant due to infection | 1 | 1
Not completed — Death | 3 | 2
Not completed — Pursue Other Treatment Options | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics and primary endpoints were calculated using the Intent-to-Treat population, which includes all subjects that underwent RNS® System implantation (191 subjects). Individuals that did not undergo initial implant (49 subjects) were withdrawn from the study and are considered screen failures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF) | Total
Number analyzed (Participants) | 97 | 94 | 191
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 6
  Between 18 and 65 years | 93 | 91 | 184
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Full Range); unit: years] | 34.0 [18 to 60] | 35.9 [18 to 66] | 34.9 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 44 | 91
  Male | 50 | 50 | 100
Duration of epilepsy [Mean (Full Range); unit: years] | 20.0 [2 to 57] | 21.0 [2 to 54] | 20.5 [2 to 57]
Number of AEDs at enrollment [Mean (Full Range); unit: number of AEDs] | 2.8 [1 to 8] | 2.9 [0 to 6] | 2.8 [0 to 8]
Mean seizure frequency [Mean (Full Range); unit: seizures/month] | 33.5 [3 to 295] | 34.9 [3 to 338] | 34.2 [3 to 338]
Seizure onset location [Number; unit: participants]
  Mesial Temporal lobe ONLY | 48 | 47 | 95
  Other | 49 | 47 | 96
Number of seizure foci [Number; unit: participants]
  Bifocal | 48 | 58 | 106
  Unifocal | 49 | 36 | 85
Prior therapeutic surgery for epilepsy [Number; unit: participants]
  Yes | 34 | 28 | 62
  No | 63 | 66 | 129
Prior EEG monitoring with intracranial electrodes [Number; unit: participants]
  Yes | 63 | 50 | 113
  No | 34 | 44 | 78
Prior vagal nerve stimulator (VNS) [Number; unit: participants]
  Yes | 30 | 34 | 64
  No | 67 | 60 | 127
Anatomical brain abnormality (by neuroimaging) [Number; unit: participants]
  Yes | 66 | 61 | 127
  No | 31 | 33 | 64
Acute benzodiazepine use (does not include daily use) [Number; unit: participants]
  Yes | 30 | 39 | 69
  No | 67 | 55 | 122

OUTCOME MEASURES:

1. Primary Outcome: Acute SAE Rate
Description: RNS® System Acute SAE Rate = the percentage of implanted subject having a serious adverse event (SAE) for the surgical implant procedure and the following month (28 days), whether reported as device-related or not.
  This outcome measure is met when the upper limit of one-sided 95% confidence interval of the observed RNS® System Acute SAE Rate does not exceed the upper limit of the one-sided 95% confidence interval of the literature-based acute SAE rate associated with the implantation of intracranial electrodes for localization procedures and epilepsy surgery combined as documented in the literature (rate = 15%; upper CI = 20%). The comparator was calculated based upon the literature, therefore the number of participants analyzed is unknown/not applicable. Referenced literature are listed within the citation section (Tanriverdi et al., 2009; Wong et al., 2009; Fountas and Smith, 2007; Hamer et al., 2002; Behrens et al., 1997).
  Primary Safety Outcome Measure was met.
Time Frame: Initial implant through 1 month post-implant
Measure: Number (95% Confidence Interval); unit: percentage of subjects with ≥ 1 SAE
Groups:
- Implanted Subjects: Subjects implanted with the RNS® System
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 191
percentage of subjects with ≥ 1 SAE | 12.0 [NA to 16.5] — The lower confidence interval is not required for this endpoint calculation.

2. Primary Outcome: Short-term Chronic SAE Rate
Description: RNS® System Short-term Chronic SAE rate = the percentage of implanted subject having a serious adverse event (SAE) for the surgical implant procedure and the following 3 months (84 days), whether reported as device-related or not.
  This outcome measure is met when the upper limit of one-sided 95% confidence interval of the observed RNS® System Short-term Chronic SAE Rate does not exceed the upper limit of the one-sided 95% confidence interval of the historical short-term chronic SAE rate for deep brain stimulation for movement disorders from the published literature (rate = 36%; upper CI = 42%). The comparator was calculated based upon the literature, therefore the number of participants analyzed is unknown/not applicable. Referenced literature are listed within the citation section (Oh et al., 2002; SSED, Activa Tremor Control System P960009; Beric et al., 2001; Behrens et al., 1997; Hariz, 2002; Joint et al., 2002; Koller et al., 2001).
  Primary Safety Outcome Measure was met.
Time Frame: Initial implant through 5 months post-implant
Measure: Number (95% Confidence Interval); unit: percentage of subjects with ≥ 1 SAE
Arm/Group | Implanted Subjects
Number analyzed (Participants) | 191
percentage of subjects with ≥ 1 SAE | 18.3 [NA to 23.4] — The lower confidence interval is not required for this endpoint calculation.

3. Primary Outcome: Change in Frequency of Disabling Seizures
Description: The outcome measure is met when a significantly greater reduction in the frequency of total disabling seizures in seen in the Treatment group when compared to the Sham group, during the Blinded Evaluation Period (BEP) relative to the Pre-Implant Period (Baseline).
  The outcome measure is the group-by-time interaction term in a generalized estimating equation (GEE), longitudinal regression model, where group refers to therapy allocation (Treatment or Sham), time refers to study period (Baseline or BEP), and the dependent variable is seizure frequency. The outcome measure was a statistically significant group-by-time interaction term, which would demonstrate a significantly greater reduction in seizure frequency in the Treatment group than the Sham group during BEP compared to Baseline Period.
  Primary Effectiveness Outcome Measure was met.
  (Note: Disabling seizures = motor simple partial seizures or complex partial seizures with or without secondarily generalized seizures.)
Time Frame: 3 months pre-implant (Baseline Period) compared to months 3, 4 and 5 post-implant (Blinded Evaluation Period)
Measure: Number (95% Confidence Interval); unit: Seizure frequency % change from Baseline
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF)
Number analyzed (Participants) | 97 | 94
Seizure frequency % change from Baseline | -37.9 [-46.7 to -27.7] | -17.3 [-29.9 to -2.3]

ADVERSE EVENTS:
Time Frame: Initial implant through 2 years post-implant
Description: SAE = a negative change in subject's physical/mental health as experienced by subject or observed by clinician, during any part of the study, that resulted in:
  * significant risks or consequences to the subject's acute or long-term health
  * serious injury or death
  * hospital admission or required invasive medical intervention to alleviate the AE
Arm/Group | Treatment Group (Stimulation ON) | Sham Group (Stimulation OFF)
Serious Adverse Events (participants affected / at risk) | 49/97 | 52/94
Other Adverse Events (participants affected / at risk) | 96/97 | 94/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (Stimulation ON) (N=97) | Sham Group (Stimulation OFF) (N=94)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acquired epileptic aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 1 (3)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angiogram cerebral (Investigations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Apraxia (Nervous system disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atonic seizures increased (Nervous system disorders) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Biopsy brain (Investigations) | 0 (0) | 1 (1)
Blindness transient (Nervous system disorders) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Complex partial seizures exacerbated (Nervous system disorders) | 1 (1) | 2 (3)
Complex partial seizures increased (Nervous system disorders) | 7 (8) | 3 (5)
Contraception (Surgical and medical procedures) | 1 (1) | 0 (0)
Conversion disorders (Psychiatric disorders) | 1 (1) | 0 (0)
Convulsive status epilepticus (Nervous system disorders) | 2 (2) | 0 (0)
Death (General disorders) | 3 (3) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 2 (2) | 2 (2)
Device lead damage (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Device lead revision (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Dysphemia (Nervous system disorders) | 0 (0) | 1 (1)
EEG monitoring (Investigations) | 8 (11) | 6 (7)
Epileptic psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1)
Hand fracture (due to seizure) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (due to seizure) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Hip fracture (due to seizure) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Implant site discharge (General disorders) | 1 (1) | 0 (0)
Implant site effusion (General disorders) | 0 (0) | 1 (1)
Implant site erosion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 4 (4) | 3 (4)
Implant site infection (due to seizure) (Infections and infestations) | 1 (1) | 1 (1)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intracranial hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (due to seizure) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (due to seizure) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Live birth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 2 (2) | 0 (0)
Medical device removal (VNS) (Surgical and medical procedures) | 2 (2) | 1 (1)
Medical observation (Investigations) | 0 (0) | 1 (2)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Nonconvulsive status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1) | 1 (1)
Premature battery depletion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Simple partial seizures (sensory) (Nervous system disorders) | 0 (0) | 1 (1)
Simple partial seizures exacerbated (motor) (Nervous system disorders) | 0 (0) | 1 (1)
Simple partial seizures increased (motor) (Nervous system disorders) | 0 (0) | 1 (1)
Simple partial seizures increased (sensory) (Nervous system disorders) | 0 (0) | 1 (1)
Skin laceration (due to seizure) (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (due to seizure) (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tendon transfer (Surgical and medical procedures) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
Thermal burn (due to seizure) (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tonic-clonic seizures exacerbated (Nervous system disorders) | 3 (3) | 4 (4)
Tonic-clonic seizures increased (Nervous system disorders) | 1 (2) | 6 (6)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Tubal ligation (Surgical and medical procedures) | 2 (2) | 0 (0)
Uterine leiomyoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (Stimulation ON) (N=97) | Sham Group (Stimulation OFF) (N=94)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (6)
Adverse drug reaction (General disorders) | 12 (17) | 18 (26)
Anxiety (Psychiatric disorders) | 6 (7) | 8 (10)
Aphasia (Nervous system disorders) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 5 (6)
Back injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (4)
Back injury (due to seizure) (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Balance disorder (Nervous system disorders) | 2 (3) | 6 (7)
Blepharospasm (Eye disorders) | 3 (3) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 7 (11)
Complex partial seizures (Nervous system disorders) | 10 (18) | 14 (17)
Complex partial seizures exacerbated (Nervous system disorders) | 7 (8) | 9 (11)
Complex partial seizures increased (Nervous system disorders) | 10 (12) | 13 (17)
Confusional state (Nervous system disorders) | 1 (2) | 8 (8)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 8 (8)
Contusion (due to seizure) (Injury, poisoning and procedural complications) | 17 (25) | 15 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 13 (16) | 14 (15)
Dermal cyst (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Device interaction (General disorders) | 4 (4) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (6)
Dizziness (Nervous system disorders) | 12 (14) | 13 (15)
Dizziness postural (Nervous system disorders) | 4 (4) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 4 (4)
Dysaesthesia (Nervous system disorders) | 9 (12) | 15 (21)
Dyskinesia (Nervous system disorders) | 3 (3) | 2 (2)
Ear infection (Infections and infestations) | 3 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Excoriation (due to seizure) (Injury, poisoning and procedural complications) | 9 (18) | 5 (7)
Eye pain (Eye disorders) | 3 (6) | 2 (2)
Fatigue (General disorders) | 11 (11) | 6 (7)
Gastroenteritis (Gastrointestinal disorders) | 3 (4) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 7 (7) | 7 (8)
Head injury (due to seizure) (Injury, poisoning and procedural complications) | 6 (7) | 10 (11)
Headache (Nervous system disorders) | 21 (28) | 27 (41)
Hypertension (Vascular disorders) | 1 (1) | 6 (6)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 0 (0)
Implant site pain (General disorders) | 41 (51) | 31 (39)
Implant site paraesthesia (General disorders) | 5 (5) | 4 (4)
Implant site swelling (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Incision site infection (Infections and infestations) | 6 (7) | 0 (0)
Influenza (Infections and infestations) | 13 (17) | 13 (19)
Insomnia (Nervous system disorders) | 8 (10) | 8 (9)
Joint injury (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Joint injury (due to seizure) (Injury, poisoning and procedural complications) | 3 (3) | 9 (10)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Limb injury (due to seizure) (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
Memory impairment (Nervous system disorders) | 8 (8) | 8 (9)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 4 (4)
Migraine (Nervous system disorders) | 3 (3) | 4 (4)
Monoparesis (Nervous system disorders) | 4 (4) | 1 (1)
Multiple injuries (due to seizure) (Injury, poisoning and procedural complications) | 4 (8) | 5 (7)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 29 (46) | 25 (40)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Nystagmus (Nervous system disorders) | 4 (4) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Pain of skin (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Panic attack (Psychiatric disorders) | 6 (7) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (5) | 8 (10)
Pharyngitis (Infections and infestations) | 2 (3) | 4 (5)
Photopsia (Nervous system disorders) | 5 (5) | 7 (8)
Polyuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Postictal state (Nervous system disorders) | 2 (2) | 4 (6)
Postoperative constipation (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Postoperative fever (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Procedural headache (Injury, poisoning and procedural complications) | 27 (30) | 27 (27)
Procedural nausea (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Pyrexia (General disorders) | 4 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (7)
Sciatica (Nervous system disorders) | 2 (2) | 3 (3)
Seasonal allergy (Immune system disorders) | 8 (8) | 3 (3)
Simple partial seizures (motor) (Nervous system disorders) | 5 (8) | 7 (12)
Simple partial seizures (sensory) (Nervous system disorders) | 11 (12) | 10 (14)
Simple partial seizures exacerbated (motor) (Nervous system disorders) | 3 (4) | 2 (2)
Simple partial seizures exacerbated (sensory) (Nervous system disorders) | 3 (5) | 2 (2)
Simple partial seizures increased (motor) (Nervous system disorders) | 3 (3) | 3 (3)
Simple partial seizures increased (sensory) (Nervous system disorders) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 4 (5) | 4 (6)
Skin laceration (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Skin laceration (due to seizure) (Injury, poisoning and procedural complications) | 18 (31) | 10 (21)
Somnolence (Nervous system disorders) | 4 (4) | 5 (5)
Swelling face (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 20 (30) | 21 (24)
Thermal burn (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 3 (5) | 2 (2)
Tongue injury (due to seizure) (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)
Tonic-clonic seizures exacerbated (Nervous system disorders) | 8 (8) | 6 (6)
Tonic-clonic seizures increased (Nervous system disorders) | 5 (7) | 8 (12)
Tooth infection (Infections and infestations) | 4 (4) | 2 (3)
Tremor (Nervous system disorders) | 8 (9) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 15 (19) | 16 (22)
Urinary tract infection (Infections and infestations) | 11 (11) | 7 (9)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Vision blurred (Eye disorders) | 4 (4) | 5 (5)
Vomiting (Gastrointestinal disorders) | 6 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each Investigator and Institution agree that the 1st publication of study results shall be a joint, multi-center publication.

Each Investigator, Coordinator, and Institution agree to submit publications to the RNS® System Study Publication Committee for review prior to submission for publication (at least 30 days for manuscripts and at least 7 days for abstracts) to assure that publication does not compromise the scientific integrity of the study or contain confidential NeuroPace information.